CLINICAL TRIAL: NCT07157501
Title: Effect of Using Aromatherapy Versus Acupressure on Pain Intensity and Sleep Pattern for Children Undergoing Abdominal Surgeries
Brief Title: Aromatherapy Versus Acupressure: Impact on Postoperative Pain and Sleep Quality in Pediatric Abdominal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Sabry Attia Hassan El malah, Dr, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAT for pain and sleep pattern
Record Dates: First submitted 2025-08-23; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Appendicitis; Hernia; Abdominal Exploration; Splenectomy
Keywords: Children; Pain; Sleep pattern; Aromatherapy; Accupressure; Abdominal surgeries
MeSH Terms: conditions — Appendicitis; Hernia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using aromatherapy for pain and sleep disturbance (Experimental): participants in this group received aromatherapy only for decreasing pain intensity and improving sleep quality for children after abdominal surgeries
  Interventions: Other: Aromatherapy inhaler
- Acupressure for pain and sleep disturbances for children after abdominal surgery (Experimental): participants in this group received acupressure for decreasing pain and improving sleep quality after abdominal surgery
  Interventions: Behavioral: Accupressure

INTERVENTIONS:
Behavioral: Accupressure — Acupressure will be applied by pressing in circular movements on the acupoint with the thumb finger first in clock wise and then anti-clock wise direction. The finger must remain at the same point on the skin and be moved in small circles
  Arms: Acupressure for pain and sleep disturbances for children after abdominal surgery
Other: Aromatherapy inhaler — The lavender inhalation application will be explained to the children and their mothers. Two drops of 100% pure organic lavender oil will poured on a cotton. The cotton will have fixed by the child at 5 cm distance from his or her nose and will asked to breathe slowly for 10-15 minutes
  Arms: Using aromatherapy for pain and sleep disturbance

SUMMARY:
The study's aim is to examine the effect of using aromatherapy versus acupressure on pain intensity and sleep pattern for children undergoing abdominal surgeries.

DETAILED DESCRIPTION:
Abdominal surgery is defined as a broad term used for various surgical procedures around the abdominal region. These can be used to treat or diagnose medical conditions present in that area. The surgery can be performed on multiple sites like the small intestines, spleen, stomach, appendix, and rectum or colon . Abdominal surgery in children can involve various techniques that depend on the organs which require an operation, that divided into two types; laparotomy and laparoscopic surgeries .

Laparotomies are defined as major surgeries which need large incisions on the abdomen of the child. These procedures require close, carful management to avoid it's major complications that extend the time of recovery. On the other hand, laparoscopic surgeries are smaller incisions made significantly than Laparotomies, that make little scars, less blood loss, decreased pain after surgery, and faster recovery . The most common cases of laparotomies among pediatric patients are adhesive bowel obstruction, adhesiolysis, open reduction of intussusception and bowel resection. While the procedures of laparoscopic surgeries that are used in pediatric patients are appendectomy, cholecystectomy, liver biopsy, ovarian distortion and orchidopexy. Pain is the serious postoperative problem that may result from operations due to tissue damage caused by surgical incisions that occurs shortly after surgery. It leads to the production of cellular breakdown and inflammatory mediators which trigger the nerve ending and send messages through the dorsal horn to the brain. The end effect of this pain transmission neuronal activity is pain perception. More than 80% of children who undergo surgical procedures experience acute postoperative pain. About 30-43% of pediatric patients report moderate or severe pain on the first postoperative day . The next most prevalent post-operative problem is insomnia. Hospitalized children frequently experience sleep disorders for many reasons such as physical condition, medications, fear of death, light, environmental noise, unpleasant odors, foreign instruments, nursing interventions, invasive procedures, complications of disease, loss of privacy and staying away from family. About 40-60% of hospitalized children have sleep disturbance . The hospitalized children stay awake for a significant amount of time; they cannot benefit from the therapeutic effects of sleep. Inadequate and unsatisfactory sleep impedes healing process by having negative effects on the immune system, wound healing process, cause fatigue, anorexia, muscle atrophy, delayed recovery, affect cognitive functions of children and increasing their level of stress and anxiety as well as, impair children's mental and physical development by directly affecting protein synthesis, cell differentiation, and growth hormone secretion .

Postoperative pain and insomnia are associated with increased morbidity and dysfunction that can delay time to ambulation and prolong the hospital length of stay. When postsurgical pain and insomnia are not appropriately managed, they may develop into chronic postoperative pain and fatigue, which, in turn, may lead to dysfunction, disability, and depression, and be difficult to manage.

Pediatric nurses play an important role in managing postoperative pain and insomnia among pediatric patients. They spend most of their time with the child and are accountable for assessment, the administration of analgesics, monitoring and reporting the outcomes of the given treatments. Some nurses believe that pain and insomnia are expected outcomes of surgery, hence, there is no need to alleviate the postoperative pain and insomnia completely .

The use of Complementary Alternative Medicine (CAM) in pediatric populations is considerably increased, especially for pain, sleep disturbance and acute conditions. The main reasons for seeking CAM were: the wish of avoiding chronic use of drugs with their related side effects, the desire of an integrated approach, the reported inefficacy of conventional medicine, and a more suitable children disposition to CAM than to pharmacological compound .

Aromatherapy is considering one type of CAM. Aromatherapy refers to the therapeutic use of essential oils absorbed through the skin or olfactory system. It's used for controlling the pain, anxiety, depression, stress, and improves the sleep pattern among pediatric patients. The benefits of lavender's aromatherapy that linalool and linalyl acetate present in this plant can stimulate parasympathetic system. In addition, linalyl acetate has narcotic effects and linalool acts as a sedative. This herb improves the heart function and as a circulatory stimulant, it has beneficial effects on coronary blood flow.

Another type of CAM is acupressure, it's a non-invasive form of traditional Chinese Medicine that is common throughout Chinese society as a method of promoting health. It includes applying of pressure manually to certain points on the body through energy pathways called meridians which spread energy in the body and connect the body parts with its organs. Appling acupressure technique can be done by using the fingertips or wristband to relieve post-operative pain and improve quality of sleep . Pain and sleep disorders are treated using both pharmacological and non-pharmacological methods. Sedative-hypnotic agents used in pharmacological treatments can reduce pain and increase the quality of sleep significantly; however, it is stated that these drugs have side effects, cause addiction and do not provide adequate sleep . Therefore, it is essential to employ and implement non-pharmacological methods that are safer and have fewer side effects than the pharmacological methods.

ELIGIBILITY:
Inclusion Criteria:

Children age 6 to 12 years of both sexes. Conscious and having a caretaker. No history of respiratory diseases or has problems with his sense of smell (for aromatherapy group).

Children undergoing abdominal surgeries such as acute appendicitis, intestinal obstruction, Inguinal and umbilical hernia

Exclusion Criteria:

Post-operative severe pain preventing children from participating in the study. Children who have chronic disease such as cardiac and renal disease. The existence of coagulation disorders, as well as skin diseases or skin burns in the pressure points where in acupressure could be applied (for acupressure group).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity as measured by the Word-Graphic Rating Scale (WGRS) | Baseline (pre-intervention), and 30 minutes post-intervention
  Pain intensity will be assessed using the Word-Graphic Rating Scale (WGRS), a validated self-report scale for children aged 6-12 years. The scale includes descriptive words along a line, ranging from "No pain" to "Worst possible pain." Children point to the word that best describes their pain level. Scores range from 0 to 10, with higher scores indicating greater pain intensity. The change from baseline to post-intervention will be analyzed.
  Unit of Measure:
  Score on a 0-10 scale
Change in sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline (pre-intervention) and at the morning of 2nd postoperative day and at the morning of 3rd postoperative day
  Pittsburgh Sleep Quality Index: It is a self-report questionnaire that assessed sleep quality and sleep pattern. The scale consists of components such as subjective sleep quality, sleep latency, habitual sleep efficiency, sleep disturbance, day time dysfunction. This rating scale consists of 30 items based on the 5 components. The scale will be used for the pre and post-test. Scoring of answer is based on 4-point rating scale (0 -3). Never - 0, Occasionally - 1, Frequently - 2, Always - 3. Scoring system : Good quality of sleep 0-30. Fair quality of sleep 31-60. Poor quality of sleep61-90

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa S.A. El Malah, PhD, Principal Investigator — Faculty of Nursing, Mansoura University
Locations (1):
- Faculty of nursing - Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No